CLINICAL TRIAL: NCT02633020
Title: A Phase 2a, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of AMG 714 in Adult Patients With Type II Refractory Celiac Disease, an In Situ Small Bowel T Cell Lymphoma
Brief Title: Study to Evaluate the Efficacy and Safety of AMG 714 in Adult Patients With Type II Refractory Celiac Disease
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CELIM-RCD-002; 2015-004063-36 (EudraCT Number)
Expanded Access: NCT03439475 (No longer available)
Record Dates: First submitted 2015-11-28; First posted 2015-12-17 (Estimated); Results first posted 2019-12-27 (Actual); Last update posted 2019-12-27 (Actual); Status verified 2019-11

CONDITIONS: Type II Refractory Celiac Disease (RCD-II); In-situ Small Bowel T-cell Lymphoma
MeSH Terms: interventions — AMG-714

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- AMG 714 (Experimental): Participants were administered 8 mg/kg AMG 714 via intravenous infusion on day 0, day 7 and every 2 weeks thereafter through week 10.
  Interventions: Biological: AMG 714
- Placebo (Placebo Comparator): Participants were administered placebo via intravenous infusion on day 0, day 7 and every 2 weeks thereafter through week 10.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: AMG 714 — Administered via a 120-minute IV infusion for a total of 7 times over 10 weeks.
  Arms: AMG 714
Biological: Placebo — Administered via a 120-minute IV infusion for a total of 7 times over 10 weeks.
  Arms: Placebo

SUMMARY:
Protocol CELIM-RCD-002 is designed to evaluate the efficacy and safety of AMG 714 for the treatment of adult patients with type II refractory celiac disease (RCD-II), an in-situ small bowel T-cell lymphoma.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed diagnosis of refractory celiac disease Type II (RCD-II)
* Greater than 20% aberrant intraepithelial lymphocytes (IEL) as assessed by flow cytometry
* On a gluten-free diet for at least 6 months
* Avoid pregnancy

Exclusion Criteria:

* Enteropathy-Associated T cell Lymphoma (EATL)
* Infections
* Immune suppression
* Clinically significant co-morbidities

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2016-04-13 (Actual); Primary Completion 2017-04-11 (Actual); Study Completion 2017-05-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amgen, MD, Study Director — Amgen
Locations (6):
- United States (2):
  - Clinical Site, San Diego, California
  - Clinical Site, New York, New York
- Clinical Site, Tampere, Finland
- Clinical Site, Paris, France
- Clinical Site, Amsterdam, Netherlands
- Clinical Site, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
Publication in peer-reviewed journals

REFERENCES:
- [Derived] Cellier C, Bouma G, van Gils T, Khater S, Malamut G, Crespo L, Collin P, Green PHR, Crowe SE, Tsuji W, Butz E, Cerf-Bensussan N, Macintyre E, Parnes JR, Leon F, Hermine O, Mulder CJ; RCD-II Study Group Investigators. Safety and efficacy of AMG 714 in patients with type 2 refractory coeliac disease: a phase 2a, randomised, double-blind, placebo-controlled, parallel-group study. Lancet Gastroenterol Hepatol. 2019 Dec;4(12):960-970. doi: 10.1016/S2468-1253(19)30265-1. Epub 2019 Sep 4. PMID 31494097
- See also: Related Info — http://www.celimmune.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 6 sites in France, Netherlands, Finland, Spain, and the United States. Participants with previously confirmed diagnosis of refractory coeliac disease (RCD) type 2 were enrolled from April 13, 2016 to January 19, 2017.
Pre-assignment Details: Participants were randomized in a 2:1 ratio to receive either 8 mg/kg AMG 714 or placebo. Randomization and initial dosing of the first 10 participants were staggered to allow observation for any possible unanticipated side effects.
Period: Overall Study
Arm/Group | AMG 714 | Placebo
Started | 19 | 9
Completed | 18 | 9
Not Completed | 1 | 0
Not completed — Adverse Event | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AMG 714 | Placebo | Total
Number analyzed (Participants) | 19 | 9 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.0 (10.2) | 68.4 (10.9) | 64.8 (10.5)
Age, Customized [Count of Participants; unit: Participants]
  18 - 64 years | 12 | 2 | 14
  65 - 84 years | 7 | 7 | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 6 | 14
  Male | 11 | 3 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 2 | 2
  Not Hispanic or Latino | 19 | 7 | 26
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 19 | 9 | 28
Percentage of Aberrant Intestinal Intraepithelial Lymphocytes (IELs) Versus Total IELs [Mean (Standard Deviation); unit: percentage of aberrant IELs] — Aberrant IELs were defined by flow cytometry as surface cluster of differentiation (CD)3-negative, intra-cellular CD3-positive IELs (sCD3-, icCD3+). Population: The per protocol (PP) population included participants who received study drug and provided evaluable data for efficacy analysis, excluded non-evaluable participants and those with major protocol deviations. Participants with atypical RCD-II were also excluded.
  percentage of aberrant IELs
    number analyzed (Participants) | 14 | 8 | 22
    (all) | 62.86 (24.889) | 57.60 (22.199) | 60.94 (23.55)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in the Percentage of Aberrant Intestinal Intraepithelial Lymphocytes With Respect to All Intraepithelial Lymphocytes
Description: The primary endpoint in this study was the change form baseline in the percentage of aberrant intestinal intraepithelial lymphocytes (IELs) with respect to total IELs, as assessed by flow cytometry (Immunological Response 1).
  Intraepithelial lymphocytes (IELS) are white blood cells interspersed between epithelial cells of the small and large intestine where they function to preserve the integrity of the mucosal barrier by protecting the epithelium against pathogen or immune-induced pathology. In refractory coeliac disease type 2, aberrant intraepithelial lymphocytes make up 20% or more of total intraepithelial lymphocytes. Aberrant IELs were defined by flow cytometry as surface cluster of differentiation (CD)3-negative, intracellular CD3-positive IELs (sCD3-, icCD3+).
Time Frame: Baseline and week 12
Population: The per protocol (PP) population included participants who received study drug and provided evaluable data for efficacy analysis, excluded non-evaluable participants and those with major protocol deviations. Participants with atypical RCD-II were also excluded from analyses of Immunological Response 1.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | AMG 714 | Placebo
Number analyzed (Participants) | 14 | 8
percent change | 2.45 (8.83) | 7.30 (11.70)
Statistical Analysis 1: Comparison: AMG 714 vs Placebo; Test type: Superiority; p = 0.7451, ANCOVA; Analysis of covariance (ANCOVA) with baseline % aberrant IELs vs total IELs as a covariate and treatment group as a fixed effect; LS Mean Difference = -4.85, 90% CI 2-sided [-30.26 to 20.56], Standard Error of Mean 14.7

2. Secondary Outcome: Percent Change From Baseline in the Percentage of Aberrant Intestinal Intraepithelial Lymphocytes With Respect to All Intestinal Epithelial Cells
Description: Percent change from baseline in the percentage of aberrant intestinal IELs with respect to intestinal epithelial cells (Immunological Response 2) is a composite endpoint calculated by multiplying the percent of aberrant IEL versus total IELs (per flow cytometry) by the percent of total IEL versus intestinal epithelial cells as assessed by immunohistochemistry.
Time Frame: Baseline and week 12
Population: The per protocol (PP) population included participants who received study drug and provided evaluable data for efficacy analysis, excluded non-evaluable participants and those with major protocol deviations. Participants with atypical RCD-II were also excluded from analyses of Immunological Response 2.
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | AMG 714 | Placebo
Number analyzed (Participants) | 14 | 8
percent change | 11.66 (15.79) | 49.88 (21.33)
Statistical Analysis 1: Comparison: AMG 714 vs Placebo; Test type: Superiority; p = 0.1803, ANCOVA; ANCOVA model with baseline % aberrant IELs vs intestinal epithelial cells as a covariate and treatment group as a fixed effect; LS Mean Difference = -38.22, 95% CI 2-sided [-95.73 to 19.29], Standard Error of Mean 27.48

3. Secondary Outcome: Percent Change From Baseline in Villous Height to Crypt Depth (VH:CD) Ratio
Description: Villi are the small fingerlike projections that line the small intestine and promote nutrient absorption and are often shortened in patients with celiac disease. Crypts are grooves between the villi that are often elongated in patients with celiac disease. A decreased VH:CD ratio indicates worsening disease and increases in the VH:CD ratio indicate an improvement in the histology of intestinal mucosa (Histological Response).
  Small bowel biopsies were performed at baseline and week 12; histological assessments were performed by a blinded central pathologist.
Time Frame: Baseline and week 12
Population: Per protocol population
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | AMG 714 | Placebo
Number analyzed (Participants) | 17 | 9
percent change | 26.44 (14.06) | 15.77 (19.36)
Statistical Analysis 1: Comparison: AMG 714 vs Placebo; Test type: Superiority; p = 0.6607, ANCOVA; ANCOVA model with baseline VH:CD ratio as a covariate and treatment group as a fixed effect; LS Mean Difference = 10.67, 95% CI 2-sided [-38.97 to 60.31], Standard Error of Mean 24.00

4. Secondary Outcome: Percentage of Participants With Improvement in Marsh Score at Week 12
Description: The Marsh classification system describes the stages of damage in the small intestine as seen under a microscope, with possible values of 0, 1, 2, 3a, 3b, or 3c. A score of 0 (best score) indicates that the intestinal lining is normal and celiac disease highly unlikely, a score of 3c (worst score) indicates increased intraepithelial lymphocytes, increased crypt hyperplasia and complete villi atrophy.
  Improvement is defined as a lower grade on the Marsh score scale compared to baseline.
Time Frame: Baseline and week 12
Population: Per protocol population
Measure: Number; unit: percentage of participants
Arm/Group | AMG 714 | Placebo
Number analyzed (Participants) | 17 | 9
percentage of participants | 35.3 | 33.3
Statistical Analysis 1: Comparison: AMG 714 vs Placebo; Test type: Superiority; p = 0.9204, Regression, Logistic; Odds Ratio (OR) = 1.09, 95% CI 2-sided [0.20 to 6.01]

5. Secondary Outcome: Percent Change From Baseline in Total Intraepithelial Lymphocyte Count at Week 12
Description: Small bowel biopsies were performed at baseline and week 12; histological assessments were performed by a blinded central pathologist. The total IEL count is the density of IELs vs intestinal epithelial cells measured by immunohistochemistry.
Time Frame: Baseline and week 12
Population: The per protocol population
Measure: Least Squares Mean (Standard Error); unit: percent change
Arm/Group | AMG 714 | Placebo
Number analyzed (Participants) | 17 | 9
percent change | 26.84 (17.90) | 39.57 (24.95)
Statistical Analysis 1: Comparison: AMG 714 vs Placebo; Test type: Superiority; p = 0.6885, ANCOVA; ANCOVA) model with baseline total IEL counts as a covariate and treatment group as a fixed effect; LS Mean Difference = -12.73, 95% CI 2-sided [-77.57 to 52.12], Standard Error of Mean 31.34

6. Secondary Outcome: Number of Weekly Bowel Movements at Baseline and Week 12
Description: Participants were asked to record every bowel movement during the study using an electronic diary. If no bowel movements were experienced by the participant on any given day, the participant was required to document this in the diary.
Time Frame: Baseline and week 12
Population: The intent-to-treat population consisted of all randomized participants who had received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: bowel movements per week
Arm/Group | AMG 714 | Placebo
Number analyzed (Participants) | 19 | 9
bowel movements per week
  Baseline: number analyzed (Participants) | 19 | 8
  Baseline | 10.3 (5.21) | 7.4 (4.03)
  Week 12: number analyzed (Participants) | 18 | 9
  Week 12 | 11.3 (5.72) | 8.3 (3.39)
Statistical Analysis 1: Comparison: AMG 714 vs Placebo; Test type: Superiority; p = 0.4469, Generalized Linear Mixed Model; Generalized linear mixed model with subject as a random effect and treatment group, time (week) and their interaction as fixed effects; Ratio of LS Means = 1.17, 95% CI 2-sided [0.77 to 1.8], Standard Error of Mean 0.24

7. Secondary Outcome: Percentage of Participants With Diarrhea at Baseline and Week 12
Description: The Bristol Stool Form Scale (BSFS) is a pictorial aid to help participants identify the shape and consistency of their bowel movements. Participants were asked to complete this form daily using an electronic diary at the time of each bowel movement. The BSFS categorizes bowel movements into 7 types, from Type 1 (separate hard lumps, like nuts; hard to pass) to Type 7 (watery, no solid pieces, entirely liquid).
  Diarrhoea was defined at least one BSFS score >= 6 for the given week.
Time Frame: Baseline and week 12
Population: Intent-to-treat population
Measure: Number; unit: percentage of participants
Arm/Group | AMG 714 | Placebo
Number analyzed (Participants) | 19 | 9
percentage of participants
  Baseline | 52.6 | 22.2
  Week 12 | 36.8 | 44.4

8. Secondary Outcome: Change From Baseline in Total Weekly Gastrointestinal Symptom Rating Scale (GSRS) Score at Week 12
Description: The GSRS is a 15-question 7-scale questionnaire used to assess 5 dimensions of gastrointestinal syndromes: diarrhea, indigestion, constipation, abdominal pain and reflux. Questions are scored between 1 (no discomfort at all) and 7 (very severe discomfort).
  The total GSRS score is calculated as the sum of the scores of all 15 questions, and ranges from 15 (no discomfort at all) to 105 (very severe discomfort in all 5 dimensions of gastrointestinal syndromes).
Time Frame: Baseline and week 12
Population: Intent-to-treat population with available data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | AMG 714 | Placebo
Number analyzed (Participants) | 18 | 8
units on a scale | -0.14 (0.13) | 0.20 (0.19)
Statistical Analysis 1: Comparison: AMG 714 vs Placebo; Test type: Superiority; p = 0.4832, Linear mixed effects repeated measures; Linear mixed effects repeated measures model with baseline value, treatment group, time point and time point-by-treatment group as fixed effects; LS Mean Difference = -0.14, 95% CI 2-sided [-0.53 to 0.26], Standard Error of Mean 0.19

9. Secondary Outcome: Change From Baseline in Total Celiac Disease GSRS (CeD-GSRS) Score at Week 12
Description: The CeD-GSRS score is derived from a subset of 10 questions from the GSRS questionnaire (questions 1, 4-9, 11, 12 and 14), which are each assessed on a scale of 1 (no discomfort at all) to 7 (very severe discomfort).
  The total CeD-GSRS score ranges from 10 (no discomfort at all) to 70 (very severe discomfort in all celiac syndromes).
Time Frame: Baseline and week 12
Population: Intent-to-treat population with available data.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | AMG 714 | Placebo
Number analyzed (Participants) | 18 | 8
units on a scale | -0.14 (0.16) | 0.17 (0.24)
Statistical Analysis 1: Comparison: AMG 714 vs Placebo; Test type: Superiority; p = 0.5561, Linear mixed effects repeated measures; Linear mixed effects repeated measures model with baseline value, treatment group, time point and a time point-by-treatment group as fixed effects; LS Mean Difference = -0.14, 95% CI 2-sided [-0.64 to 0.35], Standard Error of Mean 0.24

ADVERSE EVENTS:
Time Frame: From first dose of study drug until week 16.
Description: Other Adverse Events summarizes the non-serious occurrences of adverse events that exceed the indicated frequency threshold.
Arm/Group | AMG 714 | Placebo
All-Cause Mortality (participants affected / at risk) | 0/19 | 0/9
Serious Adverse Events (participants affected / at risk) | 5/19 | 1/9
Other Adverse Events (participants affected / at risk) | 16/19 | 8/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AMG 714 (N=19) | Placebo (N=9)
Hepatitis (Hepatobiliary disorders) | 1 | 0
Pneumococcal infection (Infections and infestations) | 1 | 0
Tuberculosis (Infections and infestations) | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 0
Cerebellar syndrome (Nervous system disorders) | 1 | 0
Peroneal nerve palsy (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AMG 714 (N=19) | Placebo (N=9)
Anaemia (Blood and lymphatic system disorders) | 2 | 0
Eosinophilia (Blood and lymphatic system disorders) | 2 | 0
Erythema of eyelid (Eye disorders) | 0 | 1
Eye swelling (Eye disorders) | 1 | 0
Visual impairment (Eye disorders) | 1 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 1
Duodenal ulcer (Gastrointestinal disorders) | 0 | 1
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Gastric ulcer (Gastrointestinal disorders) | 0 | 1
Lip dry (Gastrointestinal disorders) | 1 | 0
Lip exfoliation (Gastrointestinal disorders) | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 2 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Asthenia (General disorders) | 2 | 1
Fatigue (General disorders) | 2 | 0
Pyrexia (General disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 0 | 1
Bronchitis viral (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 1 | 0
Nasopharyngitis (Infections and infestations) | 8 | 1
Oral herpes (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 1 | 0
Respiratory tract infection (Infections and infestations) | 1 | 0
Sinusitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 2 | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase abnormal (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0
Bacterial test (Investigations) | 0 | 1
Blood albumin decreased (Investigations) | 0 | 1
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 1 | 0
Blood urine present (Investigations) | 1 | 0
Eosinophil count abnormal (Investigations) | 1 | 0
Eosinophil count increased (Investigations) | 3 | 0
Helicobacter test positive (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Prostatic specific antigen increased (Investigations) | 0 | 1
Protein total decreased (Investigations) | 0 | 1
Iron deficiency (Metabolism and nutrition disorders) | 1 | 0
Dizziness (Nervous system disorders) | 0 | 3
Dizziness postural (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 3 | 0
Paraesthesia (Nervous system disorders) | 1 | 0
Tremor (Nervous system disorders) | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 1
Sleep disorder (Psychiatric disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 1 | 0
Rosacea (Skin and subcutaneous tissue disorders) | 1 | 0
Skin plaque (Skin and subcutaneous tissue disorders) | 1 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multicenter studies, the investigator agrees not to publish any results before the first multi-center publication.

DOCUMENTS (2):
  • Study Protocol (2016-07-11): https://cdn.clinicaltrials.gov/large-docs/20/NCT02633020/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-16): https://cdn.clinicaltrials.gov/large-docs/20/NCT02633020/SAP_001.pdf